CLINICAL TRIAL: NCT02658292
Title: A Double-Blind, Randomized, Vehicle-Control, Multicenter Study to Evaluate the Efficacy and Safety of NAFT900 in Children With Tinea Capitis Aged 6 to < 13 Years
Brief Title: Safety and Efficacy of NAFT900 in Children With Tinea Capitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M902001001
Record Dates: First submitted 2016-01-12; First posted 2016-01-18 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Tinea Capitis
Keywords: fungus; antifungal; skin infection; hair infection; dermatophyte; scalp; skin; eyebrows; eyelashes; hair; Trichophyton; Microsporum; Endothrix; spores
MeSH Terms: conditions — Tinea Capitis; Cellulitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NAFT900 (Active Comparator): NAFT900 (Naftifine hydrochloride foam, 3%)
  Interventions: Drug: Naftifine hydrochloride foam, 3%
- Vehicle (Placebo Comparator): Vehicle Foam
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Naftifine hydrochloride foam, 3% — Apply NAFT900 foam twice daily to the affected area(s) plus half-inch around each affected area for 4 weeks
  Other Names: NAFT900
  Arms: NAFT900
Drug: Vehicle — Apply vehicle foam twice daily to the affected area(s) plus half-inch around each affected area for 4 weeks
  Other Names: Vehicle Foam
  Arms: Vehicle

SUMMARY:
A Double-Blind, Randomized, Vehicle-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of NAFT-900 in Children Aged 6 to < 13 Years with Tinea Capitis

DETAILED DESCRIPTION:
This is an 8-week double-blind, randomized, vehicle-controlled, multicenter study of NAFT-900 compared to vehicle in the treatment of tinea capitis in children ≥6 years to <13 years of age.

There will be approximately 60 subjects enrolled. Qualifying subjects with clinical evidence of a tinea capitis infection involving ≤ 15% of the scalp, confirmed by positive culture, will be randomized 2:1 to one of the following treatments:

* NAFT-900 (Naftifine hydrochloride foam, 3%)
* Vehicle Foam The study will consist of up to 6 visits. Subjects will apply the assigned study product twice daily to the affected area(s) for 4 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with clinical diagnosis of tinea capitis with ≤15% involvement of the scalp.
2. Subjects with positive KOH microscopy and culture [for dermatophytes].
3. Male or female subjects ≥6 years and <13 years of age on the date of the Baseline Visit.

Exclusion Criteria:

1. Subject with acute inflammatory fungal infection of the scalp (kerion)
2. Subjects with skin disease on the scalp, or any other condition or prior/present treatment which in the opinion of the investigator would interfere with the study drug's effect or assessments (e.g., psoriasis, seborrheic dermatitis).
3. Subjects who received immunosuppressant therapy, cytostatic therapy or radiation therapy within 4 weeks prior to the baseline.
4. Subjects who received systemic corticosteroids and/or systemic antibiotics within 4 weeks prior to study entry (or during study).
5. Subjects who have used systemic antifungal treatment within 4 weeks prior to the baseline.
6. Subjects who have used antifungal agents, corticosteroid preparations, ketoconazole, ciclopirox, salicylic acid, terbinafine, amorolfine, butenafine, clotrimazole, econazole, oxiconazole, sertaconazole, sulconazole, luliconazole, fluconazole, benzoic acid, griseofulvin, undecylenic acid, zinc pyrithione or selenium sulfide, or tar containing topical treatments for their scalp within 1 week prior to the baseline visit.
7. Subjects with a life-threatening condition (ex. autoimmune deficiency syndrome, cancer, unstable angina, or myocardial infarction) within the last 6 months prior to baseline visit.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Compare the proportion of subjects with complete cure | 8 weeks
  Complete cure defined as negative KOH microscopy, negative dermatophyte culture and a score of 0 on baseline signs

SECONDARY OUTCOMES:
Compare the proportion of subjects with an effective treatment | 8 weeks
  Effective treatment is defined as negative KOH microscopy, negative dermatophyte culture and a score of 0 or 1 on baseline signs
Compare the proportion of subjects with mycological cure | 8 weeks
  Mycological cure is defined as complete cure defined as negative KOH microscopy and negative dermatophyte culture

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kuligowski, MD, Study Director — Merz North America, Inc.